CLINICAL TRIAL: NCT07315672
Title: Acupressure for Cough in Lung Cancer Survivors: A Randomized Controlled Trial
Brief Title: Acupressure for Cough in Lung Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Hong Kong-Shenzhen Hospital (Other); Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW24615
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Diagnosis); Acupressure; Coughing; Symptom Cluster
Keywords: Acupressure; Cough; Lung Cancer; Dyspnea; Symptom Cluster; Symptom Burden; Fatigue; Quality of Life
MeSH Terms: conditions — Lung Neoplasms; Disease; Cough; Syndrome; Dyspnea; Fatigue | interventions — Acupressure; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (Experimental): Participants will receive an 8-week acupressure intervention. After completing two hospital training sessions, the participants will perform acupressure every day for eight consecutive weeks in their daily activities following an evidence-based acupressure protocol, which will be developed based on the Chinese meridian theory, expert consensus and a comprehensive literature review of previous evidence on LC cough management. In the first week, two training sessions will be conducted to ensure the competency of the participants in performing acupressure. Afterwards, participants will be instructed to press each of the 15 designated acupoints until they experience sensations of soreness, numbness or distension, for 1 minute per time, at least two prescribed times daily (once between 9-11 am and once between 5-7 pm), and additionally during cough episodes, wherever they feel appropriate.
  Interventions: Behavioral: acupressure
- Education (Active Comparator): Participants will receive an educational booklet that includes information on the disease and treatments of LC, causes and consequences of cough, and advice on cough prevention and management.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: acupressure — Participants will perform acupressure for 8 weeks and keep practice records in a diary log. Trainers will follow up with the participants twice weekly via phone or face-to-face to assess and reinforce their practice and address acupressure-related questions.
  Arms: Acupressure
Other: Education — Participants will receive an educational booklet in the first week after the baseline assessment and complete evaluations concurrently with the experimental group. Upon study completion, they will be offered a place on a waitlist for the same acupressure intervention provided to the experimental group.
  Arms: Education

SUMMARY:
The goal of this randomized controlled trial is to examine the effect of an acupressure intervention in alleviating cough and reducing co-occurring symptoms (dyspnea, cough, and fatigue) in patients with lung cancer.

The hypotheses are:

1. Acupressure can alleviate cough in lung cancer survivors;
2. Acupressure can reduce a cough-related symptom cluster (dyspnea-cough-fatigue) experienced by lung cancer survivors;
3. Acupressure can reduce the symptom burden and improve the health-related quality of life and functional capacity of lung cancer survivors experiencing cough.

Participants will:

Receive acupressure for 8 weeks or receive an education booklet; Keep a diary of their acupressure practice and symptoms; Be assessed at baseline (T0), early intervention (T1), post-intervention (T2), and 8 weeks after the intervention period (T3).

DETAILED DESCRIPTION:
Lung cancer survivors often exhibit multiple symptoms, among which cough and its co-occurring symptoms have been identified as a group of prevalent and persistent symptoms that substantially impact their quality of life and overall survival. Research has identified cough as the sentinel symptom of the respiratory symptom cluster in lung cancer patients, underscoring the critical need for effective management strategies. This randomized controlled trial aims to evaluate the effect of a safe and self-administerable acupressure intervention on alleviating cough, reducing the dyspnea-cough-fatigue symptom cluster, and improving symptom burden, functional capacity, and quality of life in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* have a diagnosis of LC at any stage and of any pathological type;
* have a cough symptom rating ≥3 on a 0 to 10 numeric rating scale within 7 days preceding enrollment;
* can perform acupressure independently in daily activities;
* be able to read Chinese and communicate in Cantonese or Mandarin;
* be able to provide informed consent.

Exclusion Criteria:

* have unstable chronic diseases other than LC;
* have received acupressure or acupuncture within the three months preceding study enrollment;
* have serious illnesses or other conditions that prevent the participants from following the intervention protocols;
* have a life expectancy of less than 3 months;
* Be currently participating in other research programs that may affect the outcomes under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cough | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  The cough will be evaluated using the Cough Evaluation Test (CET). The 5-item instrument assesses cough under physical, psychological and social domains, with each item graded on a five-point scale, with a higher total score indicating a greater level of symptom and an MCID of 2 points.

SECONDARY OUTCOMES:
Cough-related quality of life | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  The Mandarin Chinese version of the Leicester Cough Questionnaire (LCQ-MC) will be used to assess cough-related quality of life. The widely adopted questionnaire has established satisfactory internal consistency (with Cronbach's α between 0.74 and 0.90) and test-retest reliability (with intraclass correlation coefficients between 0.89 and 0.95). The 19-item LCQ-MC has an MCID of 3.0 points. A lower total score indicates a greater level of symptom severity and poorer cough-related quality of life.
Dyspnea-cough-fatigue symptom cluster | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  The dyspnea-cough-fatigue symptom cluster will be assessed in terms of the occurrence and severity. The presence of the symptom cluster is defined as having all three symptoms. Severity of the dyspnea-cough-fatigue symptom cluster will be quantified using the average score of all three items (dyspnea, cough, and fatigue) from the MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC).
Dyspnea | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  Dyspnea will be measured using Dyspnea-12 (D-12). The 12-item instrument consists of two subscales (physical and affective), with each item graded on a 4-point scale from 0 (no dyspnea) to 3 (severe dyspnea).
Fatigue | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  The 9-item Brief Fatigue Inventory (BFI) will be used to measure fatigue levels. The instrument has two dimensions - severity and interference, with a higher total score indicating a greater symptom burden.
Symptom burden | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  The symptom burden of the participants will be measured using the MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC), which consists of 16 symptom items and 6 interference items.
Functional capacity | Pre-intervention (T0, baseline); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  Functional capacity will be assessed using the 6-minute Walking Test (6MWT), a valid and widely used test among patients with respiratory diseases.
Health-related quality of life | Pre-intervention (T0, baseline); Early intervention (T1, 1 week after T0); Post-intervention (T2, 8 weeks after T0); Follow-up (T3, 16 weeks after T0)
  Health-related quality of life will be measured with the 36-item Functional Assessment of Cancer Therapy-Lung (FACT-L) under five dimensions: physical, emotional, social, functional well-being, and LC-specific symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Shuk Ting Cheung, PhD, Study Director — The University of Hong Kong
Locations (2):
- University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong, China
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
We are not to share IPD. All IPD will be managed confidentially, using only a unique ID for identification. Access to data is limited to the research team during the study. The principal investigator is responsible for data security.

REFERENCES:
- [Result] Luo Y, Luo J, Su Q, Yang Z, Miao J, Zhang L. Exploring Central and Bridge Symptoms in Patients with Lung Cancer: A Network Analysis. Semin Oncol Nurs. 2024 Jun;40(3):151651. doi: 10.1016/j.soncn.2024.151651. Epub 2024 May 3. PMID 38704342
- [Result] Huang WX, Xu H, Fazio SD, Vivilecchia RV. Enhancement of chiral recognition by formation of a sandwiched complex in capillary electrophoresis. J Chromatogr A. 2000 Apr 14;875(1-2):361-9. doi: 10.1016/s0021-9673(99)01166-8. PMID 10839156
- [Result] Yang X, Bai J, Zhang J, Wang Y, Zhao H, Zhu X. Symptom clusters and their impacts on the quality of life of patients with lung cancer receiving immunotherapy: A cross-sectional study. J Clin Nurs. 2025 May;34(5):1725-1740. doi: 10.1111/jocn.17321. Epub 2024 Jun 17. PMID 38886988
- [Result] Takemura N, Yorke J. Respiratory symptom cluster in people with lung cancer. Curr Opin Support Palliat Care. 2025 Jun 1;19(2):71-76. doi: 10.1097/SPC.0000000000000754. Epub 2025 Mar 19. PMID 40265563
- [Result] Molassiotis A, Vu DV, Ching SSY. The Effectiveness of Qigong in Managing a Cluster of Symptoms (Breathlessness-Fatigue-Anxiety) in Patients with Lung Cancer: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211008253. doi: 10.1177/15347354211008253. PMID 33847150
- [Result] Yorke J, Johnson MJ, Punnett G, Smith J, Blackhall F, Lloyd Williams M, Mackereth P, Haines J, Ryder D, Krishan A, Davies L, Khan A, Molassiotis A. Respiratory distress symptom intervention for non-pharmacological management of the lung cancer breathlessness-cough-fatigue symptom cluster: randomised controlled trial. BMJ Support Palliat Care. 2024 Jan 8;13(e3):e1181-e1190. doi: 10.1136/spcare-2022-003924. PMID 36283797
- [Result] Karlsson K, Olsson C, Erlandsson A, Ahlberg KM, Larsson M. Exploring Symptom Clusters and Their Measurements in Patients With Lung Cancer: A Scoping Review for Practice and Research. Oncol Nurs Forum. 2023 Oct 19;50(6):783-815. doi: 10.1188/23.ONF.783-815. PMID 37874760
- [Result] Cheville AL, Novotny PJ, Sloan JA, Basford JR, Wampfler JA, Garces YI, Jatoi A, Yang P. The value of a symptom cluster of fatigue, dyspnea, and cough in predicting clinical outcomes in lung cancer survivors. J Pain Symptom Manage. 2011 Aug;42(2):213-21. doi: 10.1016/j.jpainsymman.2010.11.005. Epub 2011 Mar 12. PMID 21398089
- [Result] Molassiotis A, Lowe M, Blackhall F, Lorigan P. A qualitative exploration of a respiratory distress symptom cluster in lung cancer: cough, breathlessness and fatigue. Lung Cancer. 2011 Jan;71(1):94-102. doi: 10.1016/j.lungcan.2010.04.002. Epub 2010 May 2. PMID 20439127
- [Result] Li Y, Wang Q, Liu C, Hu X. Symptom clusters and their impact on quality of life among Chinese patients with lung cancer: A cross-sectional study. Eur J Oncol Nurs. 2023 Dec;67:102465. doi: 10.1016/j.ejon.2023.102465. Epub 2023 Nov 7. PMID 37956567
- [Result] Chen K, Yang D, Li F, Gao L, Tian Y, Xu B, Xu X, Xu Q, Cao J. Changes in the symptom clusters of elderly patients with lung cancer over the course of postoperative rehabilitation and their correlation with frailty and quality of life: A longitudinal study. Eur J Oncol Nurs. 2023 Dec;67:102388. doi: 10.1016/j.ejon.2023.102388. Epub 2023 Jul 24. PMID 37948789